CLINICAL TRIAL: NCT04430452
Title: Phase II Trial of Durvalumab (MEDI4736) With/Without Tremelimumab for Advanced Hepatocellular Carcinoma After Palliative Hypofractionated Radiotherapy
Brief Title: Durvalumab With/Without Tremelimumab After Palliative Hypofractionated Radiotherapy for Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mary Feng, MD (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Mary Feng, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 194522; NCI-2020-03671 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Advanced Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8
Keywords: Immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; Immunoglobulin G; Disulfides; Radiation Dose Hypofractionation; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I: Durvalumab monotherapy + hypofractionated radiotherapy (RT) (Experimental): Participants undergo standard of care RT over 5 fractions once a day (QD) for 5 days. Within 3-10 days after completion of RT, participants receive durvalumab IV over 1 hour on day 1. Treatment repeats every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Radiation: Hypofractionated Radiation Therapy
- Arm II: Progression on prior programmed death-ligand 1 (PD-L1) checkpoint inhibitors (Experimental): Participants with progression on prior PD-L1 immune checkpoint inhibitor undergo standard of care hypofractionated radiotherapy (RT) over 5 fractions QD for 5 days and then receive a single, fixed dose of tremelimumab (300 mg IV) administered on Day 1, in combination with a fixed dose of durvalumab (1500 mg IV) every 28 days (+/-4 days for Cycles 2+), initiated within 3-10 days of completing RT, until confirmed radiographic progression or other criteria for discontinuation.
  Interventions: Biological: Durvalumab; Radiation: Hypofractionated Radiation Therapy; Biological: Tremelimumab
- Arm III: No previous PD-L1 checkpoint inhibitor therapy (Experimental): Participants without prior PD-L1 immune checkpoint inhibitor therapy undergo standard of care hypofractionated radiotherapy (RT) over 5 fractions QD for 5 days and then receive a single fixed dose of tremelimumab (300 mg IV) administered on Day 1, in combination with durvalumab at fixed dose of 1500 mg IV every 28 days (+/-4 days for Cycles 2+), initiated within 3-10 days of completing RT, until confirmed radiographic progression or other criteria for discontinuation.

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
  Arms: Arm I: Durvalumab monotherapy + hypofractionated radiotherapy (RT); Arm II: Progression on prior programmed death-ligand 1 (PD-L1) checkpoint inhibitors
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated RT
  Other Names: Hypofractionated Radiotherapy; hypofractionation
  Arms: Arm I: Durvalumab monotherapy + hypofractionated radiotherapy (RT); Arm II: Progression on prior programmed death-ligand 1 (PD-L1) checkpoint inhibitors
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab
  Arms: Arm II: Progression on prior programmed death-ligand 1 (PD-L1) checkpoint inhibitors

SUMMARY:
This phase II trial studies how well standard of care hypofractionated radiation therapy followed by durvalumab with or without tremelimumab works in treating patients with hepatocellular cancer (liver cancer) that has spread to other places in the body (advanced) and that is growing, spreading, or getting worse (progressing). In some patients, cancer cells and immune cells start to express signals that stop the body's immune system from killing the cancer. New drugs being developed, such as durvalumab and tremelimumab, are designed to target and block these signals and may help increase the immune response to prevent or slow down cancer growth. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may help the immune system work even better. Giving durvalumab with or without tremelimumab after radiation therapy may work better than radiation therapy alone in treating patients with liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine Objective Response Rate (ORR) (per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, excluding radiotherapy (RT)-treated lesions as targets) of Durvalumab (D), and D + Tremelimumab (T) after palliative RT in advanced Hepatocellular carcinoma (HCC) participants with or without progression on prior programmed death-ligand 1 (PD-L1) immune checkpoint inhibitor.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of study interventions.

II. Determine the efficacy of treatment interventions defined as progression-free survival (PFS), duration of response (DOR), and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. Profile peripheral blood mononuclear cell (PBMC) immune cells and plasma samples before RT, after RT, and during D or D + T immunotherapy.

II. Explore relationship between peripheral blood and PBMC immune profiles, safety/tolerability, and clinical outcomes.

III. Profile immune cells in archival pre-treatment tumor tissue for all patients and on-/post-treatment tumor samples and/or non-tumor liver tissue samples when available and explore for relationship with safety/tolerability and clinical outcomes.

IV. Determine incidence of tumor PD-L1 expression by immunohistochemistry (IHC) in pre-treatment archival tumor samples in all patients, and in on-/post-treatment tumor samples if repeat tumor sampling is obtained for clinical indications.

V. Explore relationship between tumor PD-L1 status and clinical outcomes.

VI. Explore relationship between viral hepatitis status, viral load, safety/tolerability, and clinical outcomes.

VII. Measure tumor marker alpha-fetoprotein (AFP) response to immunotherapy plus RT and explore for relationship with clinical outcomes.

VIII. Explore relationship between site of RT (liver, bone, other soft tissue), number of RT sites (1 or > 1), safety/tolerability, clinical outcomes, and changes in immune cell profiles on treatment.

OUTLINE:

All participants receive 5-fraction RT as standard treatment for symptomatic or high-risk metastases and will be sequentially assigned to treatment Arm 1. Arm 1 will be closed after the 6th patient is enrolled.

Subsequent participants will be enrolled directly into Arm 2 (progression on prior PD(L)-1 immune checkpoint inhibitor) or Arm 3 (no prior PD(L)-1 immune checkpoint inhibitor).

After completing up to 2 years of treatment, treatment for participants with ongoing clinical benefit will be decided on a case-by-case basis and follow-ed up for survival endpoints for approximately 3 years after the first treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-diagnosed HCC with progression during or after prior PD-(L)1 checkpoint inhibitor immunotherapy (e.g., nivolumab and/or pembrolizumab or atezolizumab; prior durvalumab excluded), or without prior PD-(L)1 checkpoint inhibitor immunotherapy.

   a. For patients without prior histologic or cytologic diagnosis, radiographic diagnosis is allowed provided patients meet American Association for the Study of Liver Diseases (AASLD) criteria for radiographic diagnosis.
2. At least 1 Response Evaluation Criteria in Solid Tumors (RECIST) 1.1-measurable tumor present which has not received RT or other local therapy prior to enrollment.
3. Clinical indication for RT to any site (e.g. painful primary or metastatic tumor, local complication risk such as impending biliary or vascular obstruction).
4. Child Pugh score of A, B7, or B8 provided other liver function criteria are met.
5. Eastern Cooperative Oncology Group (ECOG) 0 or 1
6. Appropriate antiviral therapy for hepatitis B virus (HBV) according to institutional standard of care with HBV deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) < 2000 IU/mL.
7. Adequate organ function as defined below:

   * Hemoglobin >= 9.0 g/dL
   * Absolute neutrophil count >= 1,200/microliter (mcL)
   * Platelet count >= 60,000/mcL
   * Serum bilirubin =< 1.5 x institutional upper limit of normal. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
   * Aspartate aminotransferase (AST) =< 2.5 x institutional upper limit of normal unless liver metastases are present in which case it can be =< 5 x upper limit of normal (ULN)
   * International normalized ratio (INR) < 1.5
   * Creatinine clearance > 30 mL/min by Cockcroft Gault formula.
8. No contraindication to immune checkpoint inhibitor immunotherapy.
9. No contraindication to RT.
10. Age >=18 years at time of study entry.
11. Life expectancy of >= 12 weeks.
12. Body weight > 30 kg (66.1 pounds).
13. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
    * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
14. Women of childbearing potential and men must agree to use adequate contraception from the time of screening through the duration of study participation and for at least 6 months after receiving combination of durvalumab plus tremelimumab and 3 months after last dose of durvalumab.
15. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
16. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the United States (US) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

1. Prior radiotherapy to tumor sites requiring RT which could compromise safety of additional treatments.
2. Prior radiotherapy to more than 30% of bone marrow or to a wide field within 4 weeks of the first study treatment.
3. Prior treatment with cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) or PD-L1 inhibitor.
4. History of allogenic organ transplantation.
5. On prior PD-1 inhibitor immunotherapy:

   * Any immune-related adverse events with National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5 grade >= 3 on any prior immunotherapy or toxicity that led to permanent discontinuation of prior immunotherapy.
   * Any AEs while receiving prior immunotherapy not resolved to grade =< 1 or resolved to baseline, with the exception of patients with endocrine AE of grade =< 2, who are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic
   * Required the use of additional immunosuppression other than corticosteroids for the management of an AE, experienced recurrence of a grade >= 3 AE if previously re-challenged, and currently require maintenance doses of > 10 mg prednisone or equivalent per day
6. Major surgery, liver-directed therapy, or any other anticancer therapy (e.g. chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) less than 4 weeks prior to enrollment
7. Any other unresolved toxicity NCI CTCAE grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

   * Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the study physician
8. Concurrent enrollment in another interventional clinical study, except only in the follow-up period of that study.
9. Participation in another interventional clinical study with an investigational product during the past 4 weeks except only in the follow-up period of that study.
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients with celiac disease controlled by diet alone
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
12. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease >= 2 years before the first dose of investigational product (IP) and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
13. History of leptomeningeal carcinomatosis.
14. History of active primary immunodeficiency.
15. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice).
16. Known human immunodeficiency virus (HIV) infection.
17. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab/tremelimumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
18. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
19. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening through the duration of study participation and for at least 6 months after receiving combination of durvalumab plus tremelimumab and 3 months after last dose of durvalumab.
20. Known allergy or hypersensitivity to IP, any of the study drugs, or any of the study drug excipients.
21. Prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
22. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
23. Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  Response is defined per Response Evaluation Criteria in Solid Tumors 1.1 as a complete response (CR) or Partial Response (PR) (CR+PR=ORR) excluding radiation therapy-treated lesions. Response will be assessed after participants complete 5 fractions of standard palliative radiotherapy (RT). Proportion of participants with a confirmed response and corresponding exact confidence intervals will be reported by Arm. Participants with unevaluable or unknown response status will be considered non-responders

SECONDARY OUTCOMES:
Proportion of participants with reported treatment-related adverse events | Up to 2 years
  The proportion of participants with reported adverse events that are determined to be definitely, possibly, or probably related to the study treatment will be reported by arm
Median Duration of overall response (DOR) | Up to 2 years
  The period measured from the time that measurement criteria are met for complete or partial response (whichever status is recorded first) until the first date that recurrent or progressive disease is objectively documented, taking as reference the smallest measurements recorded since treatment started
Median Duration of overall Complete Response (DOCR) | Up to 2 years
  The period measured from the time that measurement criteria are met for complete response (whichever status is recorded first) until the first date that recurrent or progressive disease is objectively documented, taking as reference the smallest measurements recorded since treatment started
Median Duration of overall Complete Response (DOSD) | Up to 2 years
  measurement from first dose of protocol therapy until the criteria for disease progression is met, taking as reference the smallest measurements recorded since registration. To be assigned a status of stable disease, measurements must have met the stable disease criteria at least once after study entry at a minimum interval of not less than six weeks
Median Overall survival (OS) | Up to 3 years
  Survival will be measured from the date of entry on study and from first dose of protocol therapy to the date of death due to any cause. Censoring will be performed using the date of last known contact for those who are alive at the time of analysis
Median Progression-free survival | Up to 3 years
  Progression will be calculated in months from date of first dose of protocol therapy to date of first documented radiographic and/or clinical disease progression or death from any cause. For cases without progression, follow-up will be censored at the date of last disease assessment without progression, unless death occurs within no more than 3 months following the date last known progression-free, and any death will be counted as a failure. For participants who discontinued from study for other reasons than progression or death, progression-free survival will be censored at the date last known to be progression-free.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Feng, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No